CLINICAL TRIAL: NCT03767972
Title: Energy Devices for Rejuvenation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study procedures and enrollment were stopped due to COVID-19 restrictions on non-essential research. The study was not able to continue due to change in research personnel after research was able to resume.
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Natasha Mesinkovska, Principal Investigator, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20174054
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Rejuvenation

STUDY DESIGN:
Intervention Model Description: This is a prospective clinical trial to compare various energy-based devices for the rejuvenation of the face, neck/décolletage, hands, upper and lower extremities and vagina. Adults seeking rejuvenation of either the face, neck/décolletage, hands, upper and lower extremities, trunk and/or vagina will be treated with appropriate energy-based device(s) based on investigators' discretion. If patients' require rejuvenation of multiple areas, per investigator assessment, they will be allowed to get treatment in multiple areas. Patients will be followed for 3 months post-treatment to determine if the procedure was efficacious for rejuvenation of the area(s) treated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Rejuvenation (Experimental): Adults requiring rejuvenation of either the face, neck/décolletage, hands, upper and lower extremities, trunk and/or vagina will receive energy-based treatment (Fraxel Restore, Helios III, PicoWay, Halo, ThermiVa or DiVa) based on the investigators' assessment and discretion. The treating physician will decide which energy-based device is best-suited to addressing the patients' aging concerns; although patient preference will be taken into account, ultimately the treating physician will be responsible for the correct assessment of patients' rejuvenation needs and use of appropriate energy-based devices for the final treatment.
  Interventions: Device: Energy-based device

INTERVENTIONS:
Device: Energy-based device — Patients will receive one treatment for rejuvenation using one or multiple energy-based devices based on investigator discretion.
  Other Names: Fraxel Restore, Helios III, PicoWay, Halo, ThermiVa, DiVa

SUMMARY:
Non-ablative and ablative devices are the most commonly used minimally-invasive treatments for skin rejuvenation. Current devices on the market for rejuvenation include the lasers such as the Fraxel Restore, the Halo, the Helios III, the Pico, the ThermiVa and the DiVa which have all been shown to have efficacy for the rejuvenation of the face, décolletage, hands and vagina. In this study we propose to compare the efficacy and side effect profile of these devices for skin rejuvenation of various areas of the body including the face, décolletage, hands, trunk, upper and lower extremities, and vagina.

ELIGIBILITY:
Inclusion Criteria:

1. Exhibit skin aging and will benefit from skin rejuvenation treatment of the face, neck/décolletage, trunk, hands, upper and lower extremities and/or vagina as determined by the investigator/physician.
2. Subjects between the ages of 18-85 years old, at the time of consent.
3. Subjects may be male or female.
4. Subjects with Fitzpatrick Skin type I-III (Fraxel Restore, Helios III, Pico) or I-VI (Halo, ThermiVa, DiVa).
5. Subjects must be able and willing to give written informed consent and to comply with the requirements of this protocol. The consent form has been standardized in English. For those patients who do not read and understand English, a consent form will be standardized and provided in a language that they read and understand if possible.

Exclusion Criteria:

1. Children and adolescents (less than 18 years old).
2. Subjects who are not willing or able to provide written consent.
3. Individuals with any significant medical history including skin disorders and eating disorders as determined by the investigator/physician.
4. Subjects on any substances affecting blood coagulation (including but not limited to aspirin and other non-steroid anti-inflammatory drugs, warfarin, vitamin E, fish oil, heparin, low-molecular weight heparin, novel anti-coagulants).
5. Subjects with known blood coagulopathies.
6. Subjects with a compromise of local blood supply (including but not limited to recent surgery, severe scarring, autoimmune diseases involving the face, neck/décolletage, trunk, hands or lower extremities such as lupus, morphea, sarcoid or mixed connective tissue disease) (dependent on their treatment group).
7. Subjects who have received energy-based rejuvenation treatment of the face, neck/décolletage, trunk, hands, upper and lower extremities, and/or vagina within the past 3 months (dependent on the area they are planning to treat).
8. Subjects who meet any of the contraindication criteria listed in the product information for the device the subject will be treated with.
9. Subjects who are self-reported to be currently pregnant or lactating at the time of treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Irvine, Dermatology Clinical Research Center, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rejuvenation
Started | 24
Completed | 4
Not Completed | 20

BASELINE CHARACTERISTICS:
Population: Enrollment in the clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.
Arm/Group | Rejuvenation
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 47.5 [26 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Global Aesthetic Improvement Scale - Physician
Description: Patients will be followed for post-treatment using a physician-reported 5-point likert scale (Global Aesthetic Improvement Scale) from 0="worse" to 4="very much improved".
Time Frame: 3 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rejuvenation
Number analyzed (Participants) | 4
units on a scale | 3 (0)

2. Primary Outcome: Global Aesthetic Improvement Scale - Patient
Description: Patients will be followed for post-treatment using a patient-reported 5-point likert scale (Global Aesthetic Improvement Scale) from 0="worse" to 4="very much improved".
Time Frame: 3 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rejuvenation
Number analyzed (Participants) | 4
units on a scale | 3.5 (0.58)

ADVERSE EVENTS:
Time Frame: This study includes 5 to 6 visits and takes about seven hours over a period of 6 months for all laser treatments except for PALLAS treatment. Subjects who receive treatment with the PALLAS laser will receive biweekly treatments for a total of 25 visits (including one month follow-up) and takes about 13 hours over 6 months.
Arm/Group | Rejuvenation
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03767972/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT03767972/ICF_001.pdf